CLINICAL TRIAL: NCT05767125
Title: Effect of APRV and LTV on Lung Ventilation and Perfusion in Patients With Moderate-to-severe ARDS: a Single-center, Pilot Randomized Controlled Study
Brief Title: Effect of APRV and LTV on Lung Ventilation and Perfusion in Patients With Moderate-to-severe ARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, XiaoJing Zou,MD, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUHICU202302
Record Dates: First submitted 2023-02-16; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APRV Group (Experimental): Patients with moderate-to-severe ARDS were supported with APRV.
  Interventions: Device: APRV
- LTV Group (Active Comparator): Patients with moderate-to-severe ARDS were supported with LTV.
  Interventions: Device: LTV

INTERVENTIONS:
Device: APRV — Patients with moderate-to-severe ARDS were supported with APRV.
  Arms: APRV Group
Device: LTV — Patients with moderate-to-severe ARDS were supported with LTV.
  Arms: LTV Group

SUMMARY:
Low tidal volume ventilation (LTV) has been proposed and widely used in patients with acute respiratory distress syndrome (ARDS) to prevent ventilator-induced lung injury (VILI) and mitigate its effects. The LTV strategy is intended to protect the "baby lung" from overdistension while simultaneously allowing acutely injured tissue to continually collapse. Airway pressure release ventilation (APRV) is a highly effective strategy improving lung recruitment and oxygenation in clinical studies, but its effects on lung injury and mortality is debatable. Animal studies revealed that APRV could normalize post-injury heterogeneity and reduce the risk of VILI. Our objective was to investigate the impact of APRV and LTV on regional ventilation and perfusion distribution in ARDS patients by electrical impedance tomography (EIT).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 and ≤80 years;
2. Moderate-to-severe ARDS patients according to the Berlin definition;
3. Endotracheal mechanical ventilation ≤48 h before enrollment;
4. Expected to require continuous invasive mechanical ventilation ≥72 h.

Exclusion Criteria:

1. Severe chronic obstructive pulmonary disease, severe asthma, pulmonary bulla, subcutaneous emphysema, mediastinal emphysema, etc;
2. Contraindications to the use of electrical impedance tomography (e.g., chest surgical wounds dressing or presence of pacemaker)；
3. Pulmonary interstitial lesions；
4. End-stage of chronic disease, with an expected survival period of <6 months；
5. Body mass index >35 kg/m2;
6. Refractory shock；
7. Intracranial hypertension；
8. Pregnant and parturient woman；
9. Intra-abdominal pressure persisted > 20 mmHg and could not be relieved within 24 hours；
10. Severe thoracic deformity；
11. Severe cardiac dysfunction；
12. Atrial fibrillation and other malignant arrhythmias that seriously affect cardiac output；
13. Pulmonary embolism；
14. Extracorporeal membrane oxygenation is needed；
15. Prone positioning was performed before randomization；
16. Patients who have participated in other clinical trials within 30 days；
17. Patients who have not signed informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung ventilation/perfusion matching | 24hour
  Lung ventilation/perfusion matching assessed by EIT

SECONDARY OUTCOMES:
Lung ventilation distrubution | up to 72hour
  Lung ventilation distrubution assessed by EIT
Lung perfusion distrubution | up to 72hour
  Lung perfusion distrubution assessed by EIT
Dead-space% and shunting% | up to 72hour
  Lung Dead-space% and shunting% assessed by EIT
Oxygenation index | up to 72hour
  Oxygenation index=Arterial partial pressure of oxygen /fraction of inspired oxygen
Arterial partial pressure of carbon dioxide (PaCO2) | up to 72hour
  PaCO2 is one of the key indicators of pulmonary ventilation which can be obtained from arterial blood gas analysis.
Static respiratory compliance (Crs) | up to 72hour
  Crs=tidal volume/driving pressure
Cardiac output | up to 72hour
  Cardiac output assessed by echocardiography
Right ventricular function | up to 72hour
  Right ventricular function assessed by echocardiography
Ventilator free days | up to 28days
  28d-ventilator free days after randomization
Duration of Intensive care units stay | up to 28days
  28d-duration of Intensive care units stay after randomization
Mortality after randomization | up to 28days
  28d-all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: You Shang, prof., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zou X, Zhang H, Wu Y, Li R, Gao X, Wang A, Zhao X, Yang X, Shu H, Qi H, Fu Z, Yuan S, Ma Y, Yang L, Shang Y, Zhao Z. Physiologic Comparison of Airway Pressure Release Ventilation and Low Tidal Volume Ventilation in ARDS: A Randomized Controlled Trial. Chest. 2025 Feb;167(2):453-465. doi: 10.1016/j.chest.2024.08.050. Epub 2024 Sep 17. PMID 39299389